CLINICAL TRIAL: NCT06992440
Title: Empagliflozin to Improve Right Ventricular Function in Pulmonary Arterial Hypertension
Acronym: EmPATH
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Gustavo A Heresi, MD, MS (Other)
Collaborators: The Cleveland Clinic (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Gustavo A Heresi, MD, MS, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-168; UG3HL175041 (NIH); UH3HL175041 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin (Active Comparator): Participants receive Empagliflozin 10 mg orally once daily for 24 weeks. Empagliflozin is over-encapsulated to match placebo.
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Participants receive placebo tablet over-encapsulated to match Empagliflozin orally once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10 mg tablet once daily
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — matching tablet once daily
  Arms: Placebo

SUMMARY:
Randomized, triple-masked, parallel arm clinical trial of empagliflozin versus placebo in pulmonary arterial hypertension (PAH) participants on stable approved PAH-targeted medical therapy.

DETAILED DESCRIPTION:
The central hypothesis is that treatment with empagliflozin will improve right ventricular (RV) function and other key outcomes in patients with PAH. To test this hypothesis, the EmPATH team will conduct a multicenter Phase 2 clinical trial of empagliflozin to improve right ventricular (RV) function in pulmonary arterial hypertension (PAH). Participants will be randomized in a 1:1 ratio into two arms: empagliflozin 10 mg or matching placebo orally daily for 6 months. Randomization will be stratified by enrollment site and blocked with randomly varying block sizes. The analysis plan includes no formal interim analysis of treatment efficacy or futility.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all the following criteria:

  1. Provision of signed and dated informed consent form
  2. Ability and stated willingness to comply with all study procedures and availability for the duration of the study
  3. Ability to read and write in English
  4. Male or female, aged 18 years or older, with group 1 PAH, idiopathic, heritable, associated with drugs and toxins, associated with connective tissue disease and with congenital heart disease (simple repaired or unrepaired defects) according to the current guidelines and adjudicated by the local PI
  5. PAH confirmed by right heart catheterization in the last 5 years
  6. RV dysfunction defined FAC ≤ 34.0% on echocardiography performed during the screening visit. In PVDOMICS, FAC has a strong correlation with CMR RV ejection fraction, and FAC < 34% predicts a CMR RV ejection fraction <37% with a large c-statistic of 0.9. CMR RV ejection fraction <37% is strongly associated with increased mortality and classifies PAH as high risk under the current guidelines. We do not expect this will curtail recruitment as the mean FAC in the PVDOMICS cohort is 30 ± 10%, a population like the one that will be enrolled in this study.
  7. On FDA-approved PAH-targeted therapy (any combination including infused prostacyclin analogues and sotatercept) with stable doses for at least 8 weeks or 24 weeks for sotatercept prior to the screening visit and no clinical plans to change this therapy
  8. Diuretic doses stable for at least 4 weeks prior to screening. After screening, diuretic doses may be changed as directed by the site PIs and/or the treating physician.
  9. Ability to take oral medication and willingness to adhere to the study drug regimen.
  10. For females of reproductive potential: use of highly effective contraception for at least 4 weeks prior to screening and agreement to use such a method during study participation and for an additional 2 weeks after the end of study drug administration
  11. Able to have baseline and week 24 CMR according to Imaging Core criteria, as adjudicated by the Site PI

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Current use of insulin, insulin secretagogues (sulfonylureas and meglitinides), lithium or an SGLT2 inhibitor
  2. Use of an SGLT2 inhibitor within the past 3 months prior to screening
  3. Prior documented inability to tolerate an SGLT2 inhibitor
  4. Volume depletion, as ascertained by the site PI, at screening or baseline
  5. History of diabetic ketoacidosis or type 1 diabetes mellitus
  6. Chronic alcohol or drug abuse
  7. More than one bacterial or yeast genitourinary tract infection in the year prior to enrollment
  8. Estimated glomerular filtration rate under 30 mL/minute/1.73m2 or on renal replacement therapy
  9. Pregnancy or lactation
  10. Known allergy or hypersensitivity to empagliflozin or another SGLT-2 inhibitor
  11. Currently taking or has taken another investigational drug within the past 4 weeks
  12. Enrollment in another randomized intervention trial. (Participants participating in observational trials will not be excluded).
  13. Decompensated right heart failure, as adjudicated by the site PI.
  14. Screening HbA1c >10% with symptoms such as polyuria and polydipsia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Change in RV ejection fraction measured by CMR | 24 weeks
  RV ejection fraction measured by CMR before and after treatment

SECONDARY OUTCOMES:
Change in Fractional Area Change (FAC) measured by echocardiography | 24 weeks
  Fractional Area Change (FAC) measured by echocardiography before and after treatment
Change in the 6-minute walk distance (6MWD) | 24 weeks
  6-minute walk distance (6MWD) before and after treatment
Change in plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels | 24 weeks
  NT-proBNP before and after treatment
Time to clinical worsening | 24 weeks
  Composite endpoint defined as the occurrence of death, listing for lung or heart-lung transplantation, initiation of an additional PAH-targeted medication or increase in the prostacyclin dose by ≥10% due to PAH clinical worsening judged by the treating PAH clinician, atrial septostomy, hospitalization ≥ 24 hours for worsening of PAH, or functional deterioration defined by both a worsened NYHA functional class and a decrease in 6-minute walk distance by ≥15% from baseline.
Change in Multicomponent improvement | 24 weeks
  Percentage of participants meeting all three of the following criteria at the end of the study: any improvement in NYHA class or maintenance of class I-II, increase in 6-minute walk distance by at least 30 meters, decrease in NT-proBNP by at least 30%.
Change in French risk score | 24 weeks
  Proportion of participants meeting all three low-risk criteria at the end of the study: NYHA class I or II, 6-minute walk distance > 440 meters, and NT-proBNP < 300 pg/ml at Week 24 versus baseline.
Change in health-related quality of life (HRQOL) | 24 weeks
  Change in health-related quality of life (HRQOL) using participant reported outcome:
  the Medical Outcomes Survey Short Form-36 (SF-36) instrument Physical Health Composite (PHC) score.
Change in health-related quality of life (HRQOL) | 24 weeks
  Change in health-related quality of life (HRQOL)using participant reported outcome: the PAH-specific emPHasis-10 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Heresi, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to and stored at the NHLBI BioData Catalyst (BDC) or to the data repository designated by the NHLBI when the study ends. Data and samples could be used in research. Blood samples will be stored in the EmPATH biorepository for future studies. Some of this research might take place before the EmPATH Trial close out. The research will be approved by the Steering Committee (which includes the NHLBI). At a date agreed upon with the NIH BioLINCC, the EmPATH residual blood samples accepted for storage will be shipped to BioLINCC. After the EmPATH Trial ends, members of the PAH community including members of the EmPATH Steering Committee members may request biological samples from BioLINCC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available per NIH data management
Access Criteria: Researchers can access NHLBI data and biospecimens through the BioLINCC website, requesting access to data and biospecimens in the Biorepository, and utilizing the BioData Catalyst ecosystem.